CLINICAL TRIAL: NCT01029249
Title: Oral HPV Shedding and Oral Warts After Initiation of Antiretroviral Therapy
Brief Title: Examining the Incidence of Oral Human Papillomavirus (HPV) Shedding and Oral Warts After Beginning HAART in HIV-Infected Adults
Status: Completed | Type: Observational
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTG A5272; 1U01AI068636 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and blood will be collected from participants.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ACTG A5257 participants: Participants in this study will also be enrolled in ACTG A5257.

SUMMARY:
Oral human papillomavirus (HPV) and oral warts are common health concerns for HIV-infected people. This study will examine the frequency of oral HPV DNA shedding and oral warts in HIV-infected people who are enrolled in ACTG A5257 and who are beginning treatment with highly active antiretroviral therapy (HAART).

DETAILED DESCRIPTION:
Oral HPV infection occurs at a higher rate among HIV-infected people than among the general population. Recent research in the United States and Europe has also found that HIV-infected people have a higher risk of oral and oropharyngeal squamous cell cancer than HIV-uninfected people. In one study, it was found that HPV seropositivity was associated with an increased risk of squamous cell carcinoma of the oropharynx (SCCOP). In addition to SCCOP, another HPV-related health concern is oral warts, a condition for which there is no effective treatment. Even after beginning treatment with highly active antiretroviral therapy (HAART), active HPV replication in the mouth and oropharynx may persist in HIV-infected people, leading to an increased risk of SCCOP and oral warts. The purpose of this study is to evaluate the frequency of oral HPV DNA shedding and oral warts in HIV-infected people prior to HAART initiation and at regular time points after HAART initiation.

ACTG A5257 is a study that is comparing the effectiveness of three non-nucleoside reverse transcriptase inhibitor (NNRTI)-sparing HAART regimens in treatment-naïve participants. This study will enroll participants from the ACTG A5257 study. Participants will attend a baseline study visit at the same time as their ACTG A5257 baseline study visit. At baseline and at Week 4, 16, 24, and 48 study visits, participants will undergo an examination of their mouth, throat wash and saliva collection, and behavioral questionnaires. A blood collection will also occur at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Meet inclusion criteria for and be enrolled in ACTG A5257
* Ability and willingness of participant or legal guardian/representative to provide informed consent

Exclusion Criteria:

* Co-enrollment in A5260s
* Has begun receiving HAART as part of the A5257 study
* Has ever received an HPV vaccine or plans to receive an HPV vaccine in the 6 months after study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will also be enrolled in ACTG A5257.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Type-specific oral HPV DNA shedding (presence versus absence) | Measured at baseline (measured at pre-entry and entry into A5257) and at Weeks 16 and 24
Persistence of same type HPV DNA shedding from pre-entry/baseline visits to Week 16 and 24 visits | Measured at Weeks 16 and 24

SECONDARY OUTCOMES:
Clinical diagnosis (presence versus absence) of oral warts | Measured at Weeks 16 and 24
HPV shedding at one of the pre-HAART visits | Measured at one of the pre-entry visits
CD4 count change (compared to baseline) | Measured at Weeks 4, 16, and 24
Plasma HIV-1 RNA suppression | Measured at Weeks 4, 16, and 24
Quantitative changes in HPV DNA in oral specimens obtained from participants who have the same HPV subtypes at one of the two pre-HAART visits as well as at Week 16 or 24 | Measured at Weeks 16 or 24
Clinical diagnosis (presence versus absence) or oral warts measured by a visual exam | Measured at baseline and Weeks 16, 24, and 48
Number of oral sex partners in the last month | Measured at baseline and Weeks 24 and 48
Number of oral sex partners in the last 6 months | Measured at baseline and Weeks 24 and 48
Absolute CD8 count (obtained from A5257 study data) | Measured at Weeks 0 and 24 in the A5257 study
Absolute CD4 count (obtained from A5257 study data) | Measured at Weeks 0, 24, and 48 in the A5257 study
Percentage and absolute number of CD4 cells that are interleukin (IL)-2+/interferon (IFN)+ or transforming growth factor (TGF)+ after HPV peptide stimulation measured from peripheral blood mononuclear cells (PBMCs) | Measured during the A5272 study or obtained from stored specimens
Percentage and absolute number of CD8 cells that are IFN, tumor necrosis factor (TNF), TGF+, or CD107+ after HPV peptide stimulation measured from PBMCs | Measured during the A5272 study or obtained from stored specimens
Percentage and absolute number of CD4 cells that are regulatory T cells (CD4+/CD25+/CD127low) measured from PBMCs | Measured during the A5272 study or obtained from stored specimens
Percentage of CD4 cells and CD8 cells that express CD38 and HLA-DR | Measured during the A5272 study or obtained from stored specimens
Persistence of HPV DNA of a specific type in throat wash specimens over the time course of the study | Measured during the A5272 study or obtained from stored specimens
Salivary total lgA and anti-HPV lgA and S-lgA titers | Measured during the A5272 study or obtained from stored specimens
Serum total anti-HPV lgG titers | Measured during the A5272 study or obtained from stored specimens

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Shiboski, DDS, MPH, PhD, Study Chair — Department of Orofacial Sciences, UCSF AIDS OHARA; Mark A. Jacobson, MD, Study Chair — UCSF AIDS OHARA, Positive Health Program, San Francisco General Hospital
Locations (35):
- United States (34):
  - Alabama Therapeutics CRS (5801), Birmingham, Alabama
  - University of Southern California CRS (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Stanford, Palo Alto, California
  - Ucsd, Avrc Crs (701), San Diego, California
  - University of California San Francisco AIDS CRS (801), San Francisco, California
  - University of Miami AIDS CRS (901), Miami, Florida
  - The Ponce de Leon Ctr. CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Rush University Medical Center (2702), Chicago, Illinois
  - IHV Baltimore Treatment CRS (4651), Baltimore, Maryland
  - Beth Israel Deaconess Medical Center ACTG CRS (103), Boston, Maryland
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Henry Ford Hosp. CRS (31472), Detroit, Michigan
  - Washington University CRS (2101), St Louis, Missouri
  - Cooper Univ. Hosp. CRS (31476), Camden, New Jersey
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - Cornell CRS (7804), New York, New York
  - HIV Prevention and Treatment, New York, New York
  - AIDS Care CRS (1108), Rochester, New York
  - University of Rochester ACTG CRS (1101), Rochester, New York
  - University of North Carolina AIDS CRS, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS (1601), Durham, North Carolina
  - Moses H. Cone Memorial Hosp. CRS, Greensboro, North Carolina
  - University of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - MetroHealth CRS (2503), Cleveland, Ohio
  - The Ohio State University AIDS CRS (2301), Colombus, Ohio
  - Hospital of the University of Pennsylvania CRS (6201), Philadelphia, Pennsylvania
  - The Miriam Hospital ACTG CRS (2951), Providence, Rhode Island
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS (31475), Richmond, Virginia
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- [Background] Chaturvedi AK, Engels EA, Anderson WF, Gillison ML. Incidence trends for human papillomavirus-related and -unrelated oral squamous cell carcinomas in the United States. J Clin Oncol. 2008 Feb 1;26(4):612-9. doi: 10.1200/JCO.2007.14.1713. PMID 18235120
- See also: Click here for the ACTG A5257 ClinicalTrials.gov study record. — http://clinicaltrials.gov/ct2/show/NCT00811954